CLINICAL TRIAL: NCT05540223
Title: BIOTRONIK - Safety and Clinical Performance of the Drug Eluting Resorbable Coronary Magnesium Scaffold System (Freesolve®) in the Treatment of Subjects With de Novo Lesions in Native Coronary Arteries: BIOMAG-II: A Randomized Controlled Trial
Brief Title: Safety and Clinical Performance of the Freesolve Resorbable Magnesium Scaffold System
Acronym: BIOMAG-II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C1801; BIOMAG-II - EU, Asia and AUS (Other: BIOTRONIK AG)
Record Dates: First submitted 2022-09-09; First posted 2022-09-14 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease; Atherosclerosis, Coronary; Myocardial Ischemia; Ischemic Heart Disease; Acute Coronary Syndrome; Angina Pectoris
Keywords: Resorbable Magnesium Scaffold; Sirolimus; RMS; Drug eluting absorbable metal scaffold
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Acute Coronary Syndrome; Angina Pectoris

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Freesolve RMS (Experimental): Intervention with a Freesolve Sirolimus Eluting Resorbable Coronary Magnesium Scaffold System
  Interventions: Device: Freesolve RMS
- Xience DES (Active Comparator): Intervention with a Xience Everolimus Eluting Stent System
  Interventions: Device: Xience DES

INTERVENTIONS:
Device: Freesolve RMS — Subject undergoes implantation of Freesolve RMS
  Other Names: DREAMS 3G Sirolimus Eluting Resorbable Coronary Magnesium Scaffold System
  Arms: Freesolve RMS
Device: Xience DES — Subject undergoes implantation of Xience DES
  Other Names: Xience Everolimus Eluting Stent System
  Arms: Xience DES

SUMMARY:
The objective of this study is to assess the safety and efficacy of the Freesolve in the treatment of subjects with up to two de novo lesions in native coronary arteries compared to a contemporary drug eluting stent (DES).

DETAILED DESCRIPTION:
The Biotronik BIOMAG-II clinical trial is a prospective, international, multi-center, randomized controlled, non-inferiority trial to compare the BIOTRONIK Sirolimus Eluting Resorbable Magnesium Scaffold System (Freesolve RMS) with the Xience Everolimus Eluting Stent System (Xience DES) with respect to Target Lesion Failure (TLF) rate at 12 months. A total of 1859 subjects will be enrolled at approximately 100 study sites Europe and APAC. Subjects will be randomized in a 2:1 ratio to Freesolve or Xience.

Clinical follow-up visits will take place at 1, 6, 12 and at 2-, 3-, 4- and 5-years post procedure.

ELIGIBILITY:
Clinical Inclusion Criteria:

1. Subject is ≥ 18 years and ≤ 80 years of age
2. Subject has provided written informed consent as approved by the Independent Ethical Committee (IEC) or Institutional Review Board (IRB) of the respective clinical site prior to the study related procedures
3. Subject is eligible for PCI according to the applicable guidelines
4. Subject is an acceptable candidate for coronary artery bypass surgery
5. Subjects with stable or unstable angina pectoris, documented silent ischemia/abnormal physiologic testing or hemodynamically stable non-ST elevation myocardial infarction (NSTEMI) patients without angiographic evidence of thrombus at target lesion

   Note: STEMI patients may be eligible for the study for treatment of selected non-culprit lesions, if:
   * Subject and target lesion(s) meet all inclusion and no exclusion criteria and consent occurs at least ≥ 72 hours after successful treatment of the culprit lesion(s) [lesion(s) causing the acute STEMI];
   * Subject is hemodynamically stable with documented declining cardiac biomarkers;
   * Target lesion(s) to be treated are not located in the culprit vessel(s) and are not culprit lesion(s)
6. Subject is eligible for Dual Antiplatelet Therapy (DAPT) with aspirin plus either clopidogrel, prasugrel, ticagrelor or ticlopidine
7. Documented left ventricular ejection fraction (LVEF) ≥ 30% within 6 months prior to or during the procedure (prior to randomization)
8. Subject is willing and able to comply with protocol requirements, including completion of study visits for the duration of the study

Angiographic Inclusion Criteria:

1. Subjects with a maximum of two single de novo target lesions each in separate native coronary arteries
2. Target vessel must have a reference diameter between 2.5-4.2 mm by visual estimation, which may be assisted by Quantitative Coronary Angiography (QCA) / Intravascular Ultrasound (IVUS) / Optical Coherence Tomography (OCT)
3. Target lesion must be ≤28mm in length by operator visual estimation, which may be assissted by QCA / IVUS / OCT, (or < 20 mm for target lesion(s) to be treated with a study device < 3.0 mm in diameter) and should be amenable to treatment with a single study device
4. Target lesion stenosis ≥ 50% and < 100% by operator visual estimation, which may be assisted by QCA / IVUS / OCT. Target lesion stenosis < 70% by visual estimation, should have clinical justification for treatment as per local standards.
5. Target lesion must have a Thrombolysis In Myocardial Infarction (TIMI) flow ≥1

Clinical Exclusion Criteria:

1. Subject is pregnant and/or breastfeeding or intends to become pregnant during the duration of the study
2. Subject has clinical symptoms and/or electrocardiogram (ECG) changes consistent with STEMI < 72 hours prior to the index procedure.

   Note: Hemodynamically stable non-STEMI (NSTEMI) subjects are eligible for study enrollment.
3. Subject has undergone prior PCI within the target vessel during the last 12 months prior to the index procedure or prior PCI within a non-target vessel <72 hours prior to the index procedure if successful and uncomplicated
4. Subject is on dialysis or with impaired renal function (serum creatinine > 2.5 mg/dL or 221 µmol/L, determined within 72 hours prior to the index procedure)
5. Subject has a known allergy to contrast medium that cannot be adequately premedicated, or any known allergy to aspirin, P2Y12 inhibitors, both heparin and bivalirudin, sirolimus, everolimus (or similar limus drugs), poly L-lactide, the scaffold material (magnesium, aluminium, tantalum), or Xience stent material (cobalt, chromium, tungsten, nickel, -methacrylic polymer, and fluoropolymer)
6. Subject is receiving oral or intravenous immunosuppressive therapy (inhaled steroids are permitted) or has known life-limiting immunosuppressive or autoimmune disease (e.g., human immunodeficiency virus, systemic lupus erythematosus; diabetes mellitus is permitted)
7. Life expectancy less than 1 year
8. Planned surgery or dental surgical procedure within 6 months after index procedure, unless DAPT can be maintained
9. In the investigator's opinion subject will not be able to comply with the follow-up requirements
10. Subjects under oral anticoagulation therapy (OAC) prior to index procedure unless DAPT + OAC (i.e. triple therapy) can be maintained for a minimum of 1 month
11. Subject has had a stroke or transient ischemic attack (TIA) within 6 months prior to the index procedure
12. Subject with active bleeding disorder, active coagulopathy, or any other reason, who is ineligible for DAPT
13. Subject is currently participating or plans to participate in another study with an investigational device or an investigational drug

Angiographic Exclusion Criteria:

1. Target vessel has been previously treated and the target lesion is within 5 mm proximal or distal to the previously treated lesion
2. Left main coronary artery disease
3. Target lesion was totally occluded (100% stenosis)
4. Thrombus in target vessel
5. Future planned staged PCI either in target or non-target vessel
6. Ostial target lesion within the left descending (LAD), left circumflex (LCx), or right coronary artery (within 5.0 mm of vessel origin)
7. Target lesion involves a side branch ≥ 2.0 mm in diameter that requires a two-device strategy after pre-dilatation
8. Target lesion is located in or supplied by an arterial or venous bypass graft
9. Target lesion with excessive tortuosity proximal to or within the lesion based on visual estimation or heavily calcified target lesion which cannot be adequately pre-dilated by a non-compliant and/or cutting/scoring balloon as described in angiographic exclusion criteria 10.
10. The target lesion requires treatment with the device other than the non-compliant balloon and/or cutting/scoring balloon prior to scaffold/stent placement (including but not limited to atherectomy devices, intravascular lithotripsy, drug-coated balloons etc.)
11. Target vessel was treated with brachytherapy any time prior to the index procedure.
12. Unsuccessful pre-dilatation, defined as residual stenosis > 20% (by visual estimation) and / or angiographic complications (e.g. distal embolization, side branch closure, flow-limiting dissections)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1859 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2032-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Target Lesion Failure (TLF) at 12 Months Post-Index Procedure | 12 Months
  The primary endpoint will be Target Lesion Failure (TLF) at 12 months. TLF is a composite of Cardiac Death, Target Vessel Q-wave or non-Q wave MI, or clinically driven Target Lesion Revascularization (TLR).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Haude, MD, Principal Investigator — Rheinland Klinikum Neuss GmbH Lukaskrankenhaus Neuss
Locations (1):
- Rheinland Klinikum Neuss GmbH Lukaskrankenhaus Neuss, Neuss, Germany

IPD SHARING:
Plan to Share IPD: No
An IPD plan is being developed.